CLINICAL TRIAL: NCT06810388
Title: Effect of a Family-centred Empowerment Model-based Intervention on the Caregiving Capacity and Preparedness of Caregivers of Children with Malignant Neoplasms: a Protocol for a Quasi-experimental Study
Brief Title: Impact of Family-Centered Empowerment on Caregivers of Children with Cancer: a Quasi-Experimental Study Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaowan Li (Other)
Responsible Party: Sponsor-Investigator, Xiaowan Li, Nursing, West China Second University Hospital
Organization: West China Second University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: YXKY2024460
Record Dates: First submitted 2025-01-13; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The Family-Centred Empowerment Model (FCEM) aims to empower patients and their families by defining essential elements for improving chronic care outcomes. This model builds on the Family-Centred Care philosophy, which emphasises the child's family as the "centre of capacity building"
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No interventions have been assigned to arm 'Intervention group' Intervention 'Health education inter (Experimental): This study will be divided into 2 groups, one group will implement a health education intervention program based on a family-centered empowerment model, and the other group will implement currently available care measures.And the questionnaire was completed for all patients within three days of admission, any day from three days after admission to three days before discharge, and on the day of the three days before discharge.
  Interventions: Other: Health education intervention program based on a family-centered empowerment model; Other: Implementation of routine care measures
- Routine care group (No Intervention): The control group will be offered a health education intervention program based on a family-centered empowerment model at their children next admission for chemotherapy treatment.

INTERVENTIONS:
Other: Health education intervention program based on a family-centered empowerment model — Three sessions of approximately 15-30 min each are conducted within 3 d of the child's admission to the hospital, from the fourth day to the day before discharge, and on the day before discharge. The researcher or charge nurse assesses the caregivers' mastery every week using uniform evaluation criteria and adjusts the topic or number of interventions within each phase based on mastery, with the final intervention content and timeline remaining unchanged.Health education includes: providing family caregivers of children with malignant tumors with knowledge of the disease, guidance on dietary care, instruction on how to recognize symptoms, guidance on medication, post-implantation precautions at the port of infusion, knowledge of blood markers, monitoring of the disease, and emergency treatment.
  Arms: No interventions have been assigned to arm 'Intervention group' Intervention 'Health education inter
Other: Implementation of routine care measures — Routine nursing care and current health education content will be provided, including the following: introduction to the department's environment, rules, and regulations; admission counselling; examination guidance; distribution of health education brochures; ongoing education on daily care, medication management, and health practices during hospitalisation; guidance on daily care, medication management, and health education by the nurse in charge; proactive support and communication by medical staff, including resolving questions and sharing caregiver experience; and discharge instructions with follow-up schedules for chemotherapy.
  Participants in the control group are offered an FCEM-based intervention regimen on their second admission (at the beginning of the second course of treatment), which is appropriately adapted to the control group's second chemotherapy treatment.
  Arms: No interventions have been assigned to arm 'Intervention group' Intervention 'Health education inter

SUMMARY:
The purpose of this trial is to understand the impact of a family empowerment-based intervention program on family caregivers' readiness to care and ability to care. It aims to elucidate whether a health education intervention program based on the Family Empowerment Model improves family caregivers' readiness for care and ability to care.

Participants will receive a health education program based on the family empowerment model and will complete questionnaires three days prior to admission, during hospitalization, and three days prior to discharge.This study is a non-pharmacological intervention and will not involve any changes in treatment or chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria: (1) children aged 0-18 years old, (2) those clinically diagnosed with malignant neoplasms, and (3) first-time visitors to our hospital.

Primary caregiver inclusion criteria: the caregiver is enrolled along with the child, (1) was ≥18 years of age; (2) was a member of the child's immediate family; (3) had cared for the child for the longest period among multiple caregivers; (4) had basic communication and reading skills and was proficient in Chinese; and (5) had no previous or current history of psychiatric illness or consciousness-related disorders.

Exclusion Criteria: (1)Children who abandon treatment or are transferred to a hospital while the study is in progress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Preparedness for caregiving | Completed by the patient's family caregiver, the study participant, within three days of the patient's admission to the hospital, three days after admission to three days prior to discharge, and three days before discharge
  The Caregiver Preparation Scale was used to assess parents' preparedness to care for their children.This scale consists of eight items: preparedness for physical needs, emotional needs, service planning, caregiving stress, comfort care, coping with and managing emergencies, accessing medical information resources and help, and overall caregiving preparedness. A Likert five-point scale was used, with scores ranging from zero to four, indicating "not at all prepared" to "fully prepared," and higher scores reflecting better preparedness for caregiving.
Caring capacity | Completed by the patient's family caregiver, the study participant, within three days of the patient's admission to the hospital, three days after admission to three days prior to discharge, and three days before discharge
  The Family Caregiver Task Inventory (FCTI) was used to measure and evaluate family caregivers' caregiving abilities. The FCTI is a self-assessment scale that includes five dimensions: adapting to the role of a caregiver (five items), adapting to and assisting in caregiving (five items), dealing with personal emotions (five items), adjusting to the needs of personal life and caregiving (five items), and evaluating family and social resources (five items). It consists of a total of 25 items. The FCTI uses a three-point Likert scale, with zero indicating "no difficulty," one indicating "some difficulty," and two indicating "great difficulty." Higher scores represent greater difficulty and poorer caregiving capacity.

SECONDARY OUTCOMES:
Depression Anxiety Stress | Completed by the patient's family caregiver, the study participant, within three days of the patient's admission to the hospital, three days after admission to three days prior to discharge, and three days before discharge
  The Depression Anxiety Stress Scale (DASS-21) evaluates depression, anxiety, and stress levels in family caregivers. It contains 21 items across three dimensions: depression, anxiety, and stress. The depression subscale includes items 3, 5, 10, 13, 16, 17, and 21; the anxiety subscale includes items 2, 4, 7, 9, 15, 19, and 20; and the stress subscale includes items 1, 6, 8, 11, 12, 14, and 18. A Likert four-point scale was used, with scores ranging from zero ("did not apply at all") to three ("applied most or all of the time"). Higher scores indicate higher levels of depression, anxiety, and stress.
Self-efficacy | Completed by the patient's family caregiver, the study participant, within three days of the patient's admission to the hospital, three days after admission to three days prior to discharge, and three days before discharge
  The General Self-Efficacy Scale assesses the self-efficacy of family caregivers. It contains 10 items within one dimension and is scored on a four-point Likert scale, ranging from one ("not at all true") to four ("exactly true"), with a total score of 10 to 40. Higher scores indicate better general self-efficacy.

IPD SHARING:
Plan to Share IPD: Yes
We plan to anonymize and then share the final data statistics, which will include sociodemographic information such as study participant code, age, and gender, as well as study participant readiness for care scores, ability to care scores, self-efficacy scores, and anxiety-depression scores.
Supporting Information: Analytic Code
Time Frame: We plan to anonymize and share the data after it is completed in July 2026.

REFERENCES:
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Schwarzer R, Bäßler J, Kwiatek P, et al. The assessment of optimistic self-beliefs: Comparison of the German, Spanish, and Chinese Versions of the General Self-efficacy Scale. Appl Psychol. 1997;46:69-88.
- [Background] Chan CW, Chang AM. Managing caregiver tasks among family caregivers of cancer patients in Hong Kong. J Adv Nurs. 1999 Feb;29(2):484-9. doi: 10.1046/j.1365-2648.1999.00911.x. PMID 10197950
- [Background] Clark NM, Rakowski W. Family caregivers of older adults: improving helping skills. Gerontologist. 1983 Dec;23(6):637-42. doi: 10.1093/geront/23.6.637. No abstract available. PMID 6662379
- [Background] Liu Y, Wang M, Dong X. Reliability and validity of Chinese Version of the Caregiver Preparedness Scale in caregivers of stroke survivors. Chin J Prac Nuts. 2016;32:1045-8.
- [Background] Archbold PG, Stewart BJ, Greenlick MR, Harvath T. Mutuality and preparedness as predictors of caregiver role strain. Res Nurs Health. 1990 Dec;13(6):375-84. doi: 10.1002/nur.4770130605. PMID 2270302
- [Background] Alhani F. Design and evaluation of family-centered empowerment model to prevent iron deficiency anemia. Tehran: Tarbiat Modarres University. Published online; 2003.
- [Background] Alhani F, Asghari-Jafarabadi M, Norouzadeh R, Rahimi-Bashar F, Vahedian-Azimi A, Jamialahmadi T, Sahebkar A. The effect of family-centered empowerment model on the quality of life of adults with chronic diseases: An updated systematic review and meta-analysis. J Affect Disord. 2022 Nov 1;316:140-147. doi: 10.1016/j.jad.2022.07.066. Epub 2022 Aug 11. PMID 35964767
- [Derived] Li X, Yang Y, Chen Q, Ma J, Lu F, Luo X. Effect of a Family-Centered Empowerment Model-Based Intervention on the Caregiving Capacity and Preparedness of Caregivers of Children With Malignant Neoplasms: Protocol for a Quasi-Experimental Study. JMIR Res Protoc. 2025 Jul 29;14:e73304. doi: 10.2196/73304. PMID 40729689